CLINICAL TRIAL: NCT00282477
Title: Prospective Controlled Trial to Evaluate Erectile Function, Fertility and Sperm Count in Male Cyclists Compared to Age Matched Controls
Brief Title: Trial to Evaluate Erectile Function, Fertility and Sperm Count in Male Cyclists Compared to Age Matched Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-4031-IM-CTIL
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Erectile Dysfunction; Azoospermia
Keywords: cyclist
MeSH Terms: conditions — Erectile Dysfunction; Azoospermia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Bicycle riding is associated with related diverse urogenital symptoms ranging from genital numbness to erectile dysfunction (ED). Very little is known about the quality of sperm in cyclists and whether a connection exists between erectile dysfunction and azoospermia.

ELIGIBILITY:
Inclusion Criteria:

* Males ages 20-35, with at least 2 years of bicycle riding, at least 2 hours a week.

Exclusion Criteria:

* History of prostatic surgery, testicular surgery, or single testis,
* Patients after chemotherapy,
* Patients receiving hormonal therapy,
* Patients receiving alpha blockers for any indication.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Igael Madgar, M.D, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel